CLINICAL TRIAL: NCT04526925
Title: A Physiologic Research to Assess the Effect of an Inline Filter During Cardiopulmonary Exercise Testing (CPET): A Healthy Volunteer Study
Brief Title: The Effects of Filter During CPET on WOB and Aerosol Particle Concentrations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Staffing issues
Sponsor: Rush University Medical Center (Other)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CPET-001
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Transmission, Patient-Professional
Keywords: CardioPulmonary Exercise Testing; Aerosol Particle Size Distribution; Physiologic Responses; Filter

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- standard CPET (Active Comparator): Standard CPET will be performed without in-line filter
  Interventions: Other: Standard mouthpiece
- standard CPET with in-line filter (Experimental): An in-line filter will be placed on the mouthpiece during standard CPET
  Interventions: Device: Respiratory filter in-line placed with the standard mouthpiece

INTERVENTIONS:
Device: Respiratory filter in-line placed with the standard mouthpiece — The respiratory filter is a device that removes solid/large particles from gas
  Arms: standard CPET with in-line filter
Other: Standard mouthpiece — The mouthpiece is the interface that is placed on participant's face in order to measure all the breathing physilogic responses
  Arms: standard CPET

SUMMARY:
Due to the concerns of virus transmission during COVID-19 pandemic, multiple respiratory societies postpone or limit pulmonary function test, especially cardiopulmonary exercise test (CPET), as patients may generate large amount of aerosol particles during test but it is conventionally performed without filter. This study aims to investigate the effects of reducing aerosol particle concentrations in the room air during CPET by placing an inline filter, and to assess the effects of filter on the physiologic responses during CPET.

DETAILED DESCRIPTION:
The subject will spend two visits one hour each day (~ 1 hour) in the PFT lab and will have two separate CPET (Vmax Encore PFT System, Vyaire medical, Mettawa, IL) tests performed by registered pulmonary function technologists. One day the test will be performed with the inline filter during CPET, and the second day the CPET will be performed without a filter. During the test, electrocardiogram (ECG) electrodes will be attached to participants as well as a mask, and their heart rate will be measured for 10 minutes at rest, and then they will ride bicycle for 20 minutes at different levels of intensity. The work rate increment will be the same for both tests. All gas exchange and aerosol particle concentrations measures will be compared with Bland Altman analysis and paired t-testing.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65, Male or Female
* Normal exercise tolerance without dyspnea or clinically important limitation of exercise tolerance.

Exclusion Criteria:

* Complicated heart or lung disease
* Pregnancy
* Complex arrhythmias
* Severe Anemia
* Uncontrolled Diabetes, hypertension, or untreated thyroid disease
* Has any of the following symptoms in the last 21 days: sore throat, cough, chills, body aches for unknown reasons, shortness of breath for unknown reasons, loss of smell, loss of taste, fever at or greater than 100 degrees Fahrenheit.
* COVID-19 test positive within 21 days.
* Any Disease that the PI feels will markedly increase the risk of CPET testing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-29 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Li, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared

REFERENCES:
- [Background] Li J, Fink JB, Ehrmann S. High-flow nasal cannula for COVID-19 patients: low risk of bio-aerosol dispersion. Eur Respir J. 2020 May 14;55(5):2000892. doi: 10.1183/13993003.00892-2020. Print 2020 May. PMID 32299867
- [Background] Dhand R, Li J. Coughs and Sneezes: Their Role in Transmission of Respiratory Viral Infections, Including SARS-CoV-2. Am J Respir Crit Care Med. 2020 Sep 1;202(5):651-659. doi: 10.1164/rccm.202004-1263PP. No abstract available. PMID 32543913
- [Background] Hull JH, Lloyd JK, Cooper BG. Lung function testing in the COVID-19 endemic. Lancet Respir Med. 2020 Jul;8(7):666-667. doi: 10.1016/S2213-2600(20)30246-0. Epub 2020 May 29. No abstract available. PMID 32479795
- [Background] Gemicioglu B, Borekci S, Dilektasli AG, Ulubay G, Azap O, Saryal S. Turkish Thoracic Society Experts Consensus Report: Recommendations for Pulmonary Function Tests During and After COVID 19 Pandemic. Turk Thorac J. 2020 May;21(3):193-200. doi: 10.5152/TurkThoracJ.2020.20107. PMID 32584237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized crossover study, all the 10 participants performed cardiopulmonary exercise test (CPET). During the test, they will be randomly assigned to Standard CPET Without Filter first, then Standard CPET With Filter, or Standard CPET With Filter first, then Standard CPET Without Filter. The time period between two tests were 48 hours.
Groups:
- CPET Without a Filter First Then CPET With a Filter: Standard CPET will be performed without an in-line filter first then CPET will be performed with an in-line filter
  The filter is connected to the mouthpiece during CPET
- CPET With a Filter First Then CPET Without a Filter: Standard CPET will be performed with an in-line filter first then CPET will be performed without an in-line filter
Period: First Intervention
Arm/Group | CPET Without a Filter First Then CPET With a Filter | CPET With a Filter First Then CPET Without a Filter
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | CPET Without a Filter First Then CPET With a Filter | CPET With a Filter First Then CPET Without a Filter
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CPET Without a Filter First Then CPET With a Filter: Standard CPET will be performed without an inline filter first then CPET will be performed with an inline filter.
- CPET With a Filter First Then CPET Without a Filter: Standard CPET will be performed with an inline filter first then CPET will be performed without an inline filter.
- Total: Total of all reporting groups
Arm/Group | CPET Without a Filter First Then CPET With a Filter | CPET With a Filter First Then CPET Without a Filter | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (7.4) | 32.8 (9.2) | 32.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 3 | 5
  Asian | 2 | 2 | 4
  Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Peak Aerosol Particle Concentrations During CPET With a Filter and Without a Filter
Description: The peak aerosol particle concentrations between the situations with and without an in-line filter are reported. The peak concentrations of aerosol particles generated by subjects during CPET, are measured as particles per cubic centimeters of room air. The device measured the concentrations every 6 seconds, it continuously recorded the data for 45 minutes since CPET started and peak concentrations were reported.
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: particles per cubic centimeters
Arm/Group | Standard CPET | Standard CPET With In-line Filter
Number analyzed (Participants) | 10 | 10
particles per cubic centimeters | 204.3 (50.6) | 197.1 (4.6)

2. Primary Outcome: The Peak Minute Ventilation With and Without a Filter
Description: During CPET, participants' breathing volume (minute ventilation) is continuously monitored. The peak minute ventilation with and without a filter is reported.
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: liter per minute
Arm/Group | Standard CPET | Standard CPET With In-line Filter
Number analyzed (Participants) | 10 | 10
liter per minute | 86.1 (22.7) | 88.1 (21.8)

3. Primary Outcome: The Peak Oxygen Uptake With and Without a Filter
Description: During CPET, participants' oxygen consumption (namely, oxygen uptake) is continuously monitored. The peak oxygen uptake with and without an inline filter are reported.
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: liter per minute
Arm/Group | Standard CPET | Standard CPET With In-line Filter
Number analyzed (Participants) | 10 | 10
liter per minute | 2.37 (0.75) | 2.42 (0.75)

4. Primary Outcome: The Peak Carbon Dioxide Output With and Without a Filter
Description: During CPET, participants' exhaled volume of carbon dioxide (CO2) (namely, CO2 output) is continuously monitored. The peak CO2 output with and without an inline filter are reported.
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: liter per minute
Arm/Group | Standard CPET | Standard CPET With In-line Filter
Number analyzed (Participants) | 10 | 10
liter per minute | 2.84 (0.85) | 2.80 (0.80)

5. Secondary Outcome: The Peak Heart Rate With and Without a Filter
Description: During CPET, patients' heart rate is continuously monitored, and the peak heart rate with and without an inline filter are reported.
Time Frame: 45 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Standard CPET | Standard CPET With In-line Filter
Number analyzed (Participants) | 10 | 10
beats per minute | 164.7 (11.1) | 167.1 (9.2)

ADVERSE EVENTS:
Time Frame: 1 hour
Description: Cardiac arrest or death
Arm/Group | Standard CPET | Standard CPET With In-line Filter
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT04526925/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT04526925/ICF_001.pdf